CLINICAL TRIAL: NCT06284356
Title: Pan Immune Inflammation Value for Determining Perioperative Complications of Laparoscopic Sleeve Gastrectomy: A Prospective Cohort Study
Brief Title: Pan Immune Inflammation Value for Perioperative Complications of Laparoscopic Sleeve Gastrectomy
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Collaborators: Elazig Special Eastern Anatolian Hospital (Unknown)
Responsible Party: Principal Investigator, Mehmet Buğra Bozan, Professor, Associate, Kahramanmaras Sutcu Imam University
Other Study IDs: IRB Session 2022/14 Protocol 6
Record Dates: First submitted 2024-01-20; First posted 2024-02-28 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Morbid Obesity; Laparoscopic Sleeve Gastrectomy; Post Operative Complicaiton
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients without complications after LSG
  Interventions: Procedure: Laparoscopic Sleeve Gastrectomy
- Patients with complications after LSG
  Interventions: Procedure: Laparoscopic Sleeve Gastrectomy
- Control Group

INTERVENTIONS:
Procedure: Laparoscopic Sleeve Gastrectomy — Laparoscopic Sleeve Gastrectomy
  Groups: Patients with complications after LSG; Patients without complications after LSG

SUMMARY:
Morbid obesity emerges as a problem that causes serious complications and increased mortality rates. The most effective treatment for morbid obesity today is surgical treatment. The most preferred type of surgery in morbid obesity surgery in Turkey and around the world is Laparoscopic Sleeve Gastrectomy (LSG).

While postoperative complications are divided into early and late complications, complications that develop during surgery and in the postoperative period before discharge are defined as perioperative complications. Early surgical complications after LSG include complications such as staple line bleeding, leaks, pulmonary thromboembolism, and torsion of the remnant stomach. It is important to detect these complications, which can be controlled with early intervention in the perioperative period.

Monitoring blood parameters and monitoring inflammation are methods that are easily accessible and provide rapid evaluation. Platelet lymphocyte ratio (PLR) and neutrophil-lymphocyte ratio (NLR), which are used in the evaluation and detection of postoperative complications, have shed light on studies in this direction. Pan immune inflammation value (PIV) is calculated from blood parameters and has been used to evaluate prognosis and chemotherapy results in colorectal cancer.

In this study, the diagnostic importance of changes in NLR, PLR, and PIV values in the preoperative and postoperative periods will be investigated in detecting complications that develop in the perioperative period before discharge in patients who underwent LSG.

DETAILED DESCRIPTION:
Patients who will undergo LSG due to morbid obesity will be included in the study. Patients who are completely healthy, not morbidly obese, and have no additional disease will be taken as the control group. Reference range values will be obtained by taking a complete blood count from the control group once. From patients who will undergo LSG, routine pre-operative complete blood count values, and postoperative 24th-hour complete blood count values will be taken. PLR, NLR, and PIV will be calculated manually from these complete blood count samples and the change in these parameters will be evaluated between patients who develop complications and those who do not.

In descriptive statistics, categorical data will be given as number (n) and percentage (%). Numerical data will be given as mean ± standard deviation (SD) (minimum-maximum data) or median (25% - 75% values) depending on their compliance with normal distribution. The Kolmogorov-Simirnov test will be used to determine the distribution of normality. A p-value <0.05 is accepted as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Completely normal, healthy individuals with no additional diseases and BMI values of 19-24 kg/m2 for the control group
* Older than 18 years who will undergo Laparoscopic Sleeve Gastrectomy
* Patients with a body mass index (BMI) value ≥ 40 kg/m2 and no known comorbidities
* Patients with a BMI value ≥ 35 kg/m2 and additional comorbid diseases (such as Diabetes, Hypertension, Asthma, and Chronic Obstructive Pulmonary Disease)

Exclusion Criteria:

* Individuals under 18 years of age and morbid obesity patients
* Patients who indicate elective surgery due to morbid obesity and who are planning for non-LSG morbid obesity surgery
* Patients who do not want to participate in the study
* Patients with additional diseases such as concurrent malignancy or rheumatological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Morbid Obesity cases preparing for LSG
  * Patients with a body mass index (BMI) value ≥ 40 kg/m2 and no known comorbidities
  * Patients with a BMI value ≥ 35 kg/m2 and additional comorbid diseases (such as Diabetes, Hypertension, Asthma, and Chronic Obstructive Pulmonary Disease)
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Complication prediction after LSG with complete blood cell parameters | 2022-2023
  Blood sample changes after LSG with complete blood cell parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaras SIU, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kirkil C, Aygen E, Korkmaz MF, Bozan MB. QUALITY OF LIFE AFTER LAPAROSCOPIC SLEEVE GASTRECTOMY USING BAROS SYSTEM. Arq Bras Cir Dig. 2018 Aug 16;31(3):e1385. doi: 10.1590/0102-672020180001e1385. PMID 30133677
- [Background] Bozan MB, Kutluer N, Aksu A, Bozan AA, Kanat BH, Boyuk A. IS BODY MASS INDEX AND OBESITY SURGERY MORTALITY SCORE IMPORTANT IN PERIOPERATIVE COMPLICATIONS OF LAPAROSCOPIC SLEEVE GASTRECTOMY BEFORE DISCHARGE? Arq Bras Cir Dig. 2021 Oct 15;34(2):e1602. doi: 10.1590/0102-672020210002e1602. eCollection 2021. PMID 34669891
- [Background] Bozan MB. Gall Bladder Stone Formation in the Postoperative First Year After Sleeve Gastrectomy. Laparosc Endosc Surg Sci. 2020;27(1):25-9
- [Background] Dogan F, Dincer M. Mini-gastric Bypass Complications and the Value of the Preoperative Neutrophil to Lymphocyte Ratio in Early Prediction of Complications. J Coll Physicians Surg Pak. 2021 Jan;31(1):70-73. doi: 10.29271/jcpsp.2021.01.70. PMID 33546537
- [Background] Ortiz-Lopez D, Acosta-Merida MA, Casimiro-Perez JA, Silvestre-Rodriguez J, Marchena-Gomez J. First day postoperative values of the neutrophil-to-lymphocyte ratio, platelet-to-lymphocyte ratio, and C-reactive protein as complication predictors following gastric oncologic surgery. Rev Gastroenterol Mex (Engl Ed). 2022 Apr-Jun;87(2):142-148. doi: 10.1016/j.rgmxen.2021.11.003. Epub 2021 Nov 15. PMID 34794921
- [Background] Gambichler T, Said S, Abu Rached N, Scheel CH, Susok L, Stranzenbach R, Becker JC. Pan-immune-inflammation value independently predicts disease recurrence in patients with Merkel cell carcinoma. J Cancer Res Clin Oncol. 2022 Nov;148(11):3183-3189. doi: 10.1007/s00432-022-03929-y. Epub 2022 Jan 31. PMID 35098389
- [Background] Sato S, Shimizu T, Ishizuka M, Suda K, Shibuya N, Hachiya H, Iso Y, Takagi K, Aoki T, Kubota K. The preoperative pan-immune-inflammation value is a novel prognostic predictor for with stage I-III colorectal cancer patients undergoing surgery. Surg Today. 2022 Aug;52(8):1160-1169. doi: 10.1007/s00595-021-02448-6. Epub 2022 Jan 11. PMID 35015151